CLINICAL TRIAL: NCT02853903
Title: Comparison of Autogenic and Allogenic NK Immunotherapy on the Outcome of Recurrent Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Auto-allo NK
Record Dates: First submitted 2016-07-28; First posted 2016-08-03 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2018-07

CONDITIONS: Malignant Solid Tumour
Keywords: solid tumor; NK immunotherapy

ARMS (2):
- Allogenic NK immunotherapy (Experimental): In this group, the patients will receive more than 4 times of allogenic NK immunotherapies in 3 months. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Biological: NK immunotherapy
- Autogenic NK immunotherapy (Active Comparator): In this group, the patients will receive more than 4 times of autogenic NK immunotherapies in 3 months. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Biological: NK immunotherapy

INTERVENTIONS:
Biological: NK immunotherapy — Each treatment: 8-10 billion cells in all, transfusion in 3 times, i.v.

SUMMARY:
The aim of this study is the efficacy of autogenic and allogenic natural killer (NK) immunotherapy on recurrent solid tumors.

DETAILED DESCRIPTION:
By enrolling patients with multiple kinds of solid tumor adapted to enrolled criteria, this study will document for the first time the short/long term efficacy of auto/allogenic NK cells.The outcome will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 5 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Relief degree of tumors | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
Overall survival（OS） | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, MD, PhD, Principal Investigator — Fuda Cancer Hospital, Guangzhou
Locations (1):
- Fuda cancer institute of Fuda cancer hospital, Guangzhou, Guangdong, China